CLINICAL TRIAL: NCT06902688
Title: Timely Ordering of Pharmacogenetic Testing in Pediatric Oncology
Brief Title: Timely Ordering of Pharmacogenetic Testing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lillian Sung, Chief Clinical Data Scientist, Paediatric Oncologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 3423
Record Dates: First submitted 2025-03-13; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-02

CONDITIONS: Machine Learning; Prediction Models; Pediatrics; Precision Medicine
Keywords: precision medicine; machine learning; pharmacogenetics; prediction models; pediatrics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ML model (Experimental): Participants predicted by an ML model to receive a "targeted medication" within three months following admission.
  Interventions: Other: ML-based intervention

INTERVENTIONS:
Other: ML-based intervention — A ML-based model will predict and identify participants that are at high-risk of receiving a targeted medication within three months after their hospital admission date.

SUMMARY:
The goal of this trial is to learn if a machine learning (ML) model can help optimize drug therapy in the pediatric population. The main question[s] it aims to answer are whether a machine learning model predicting receipt of a targeted medication within the next three months:

* Increases the offering of pharmacogenetic testing prior to receipt of a targeted medication
* Increases the number of patients with pharmacogenetic results prior to receipt of a targeted medication
* Increases the number of patients who have alteration in medication choice or dose based on pharmacogenetic results

This trial only focuses on the prediction and provision of participants with a high-risk of receiving a medication with a pharmacogenetic indication in the next three months.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of a ML model in predicting patients at high risk of requiring a "targeted medication" within the next three months. A machine learning model will predict, the morning following admission to any inpatient service, whether there will be receipt of a targeted medication within the next three months. The research team will be notified regarding eligible patients each morning, and the research team or pharmacogenomics team will approach the patient's primary care team as applicable. By leveraging ML, this study seeks to enhance the identification of patients who would benefit from such medications in a timely and resource-efficient manner.

The study team identified specific medications as indications for pharmacogenetic testing based on prevalence and level of evidence for modifying prescribing practices. These pre-selected medications are referred to as "targeted medications" and are as follows: azathioprine, brivaracetam, clobazam, clopidogrel, flecainide, phenytoin, tacrolimus, voriconazole and warfarin. Only systemically administered (oral, subcutaneous, intramuscular or intravenous) medications or prescriptions (e.g. not topical, intrathecal or intravitreal) are included. Phenytoin was only considered if given orally (to exclude emergency administration without a plan for ongoing treatment).

Pharmacogenetic testing will be offered to participants and conducted as addressed in an associated pharmacogenetic testing protocol (REB# 1000053445 PI: Iris Cohn).

ELIGIBILITY:
Inclusion Criteria:

* Inpatient at The Hospital for Sick Children
* Between 6 months to 18 years old

Exclusion Criteria:

* Prior pharmacogenetic testing and/or prior receipt of a targeted medication
* Current Intensive Care Unit (ICU) admission
* Expected hospital discharge is prior to midnight on the day of admission

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 275 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients with Pharmacogenetic Testing | Day 1 to 3 months
  The primary outcome will be the proportion of patients with pharmacogenetic testing offered among those who receive a medication with a pharmacogenetic indication within three months of prediction time. Testing must be offered prior to receipt of the first targeted medication.

SECONDARY OUTCOMES:
Number of patients with pharmacogenetic results available prior to receipt of targeted medication | Day 1
  Measured via chart review
Number of patients who have alteration in medication choice or dose based on pharmacogenetic results | Day 1
  Measured via chart review

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Sung, MD, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No